CLINICAL TRIAL: NCT04997265
Title: Strategies for Anticoagulation During Venovenous ECMO: The SAFE-ECMO Pilot Trial
Brief Title: Strategies for Anticoagulation During Venovenous ECMO
Acronym: SAFE-ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Whitney Gannon, Acute Care Nurse Practitioner, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202210
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Hypoxemic Respiratory Failure; Anticoagulant-induced Bleeding; Thromboembolism
Keywords: ARDS; Hypoxemic respiratory failure; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Respiratory Insufficiency; Thromboembolism

STUDY DESIGN:
Intervention Model Description: Single center, open-label, parallel-group, randomized pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Anticoagulation (Experimental): For patients assigned to the low intensity anticoagulation strategy, clinical teams will be instructed to initiate low intensity anticoagulation at doses and frequencies commonly used for deep vein thrombosis (DVT) prophylaxis. The choice of anticoagulant, dose, and frequency of administration will be deferred to treating clinicians.
  Interventions: Other: Low intensity anticoagulation
- Moderate Intensity Anticoagulation (Active Comparator): For patients assigned to the moderate intensity anticoagulation group, clinical teams will be instructed to initiate a continuous infusion of moderate intensity anticoagulation targeting either a partial thromboplastin time (PTT) of 40-60 seconds or an Anti-Xa level of 0.2 to 0.3 IU/mL. The choice of anticoagulant and approach to dosing will be deferred to treating clinicians.
  Interventions: Other: Moderate Intensity Anticoagulation

INTERVENTIONS:
Other: Low intensity anticoagulation — Participants assigned to the low intensity anticoagulation strategy will receive anticoagulation at doses used for DVT prophylaxis in critically ill patients. The choice of agent (e.g. heparin or enoxaparin) and specific dosing will be at the discretion of the treating clinicians and will be prospectively recorded.
  Arms: Low Intensity Anticoagulation
Other: Moderate Intensity Anticoagulation — Patients assigned to the moderate intensity anticoagulation strategy will receive anticoagulation targeting a PTT goal of 40-60 seconds or anti-Xa level of 0.2 to 0.3 IU/mL. Choice of anticoagulant and monitoring strategy (PTT or anti-Xa level) will be at the discretion of the treating clinicians and will be prospectively recorded. Anticoagulant drips will be titrated according to institutional protocols. For patients who survive to decannulation, the infusion will be stopped one hour prior to decannulation.
  This approach to anticoagulation reflects the current approach for patients receiving V-V ECMO at Vanderbilt University Medical Center and is similar to protocols widely adopted for patients receiving V-V ECMO at other centers.
  Arms: Moderate Intensity Anticoagulation

SUMMARY:
Moderate intensity titrated dose anticoagulation has been used in patients receiving extracorporeal membrane oxygenation (ECMO) to prevent thromboembolism and thrombotic mechanical complications. As technology has improved, however, the incidence of thromboembolic events has decreased, leading to re-evaluation of the risks of anticoagulation, particularly during venovenous (V-V) ECMO. Recent data suggest that bleeding complications during V-V ECMO may be more strongly associated with mortality than thromboembolic complications, and case series have suggested that V-V ECMO can be safely performed without moderate or high intensity anticoagulation. At present, there is significant variability between institutions in the approach to anticoagulation during V-V ECMO. A definitive randomized controlled trial is needed to compare the effects of a low intensity fixed dose anticoagulation (low intensity) versus moderate intensity titrated dose anticoagulation (moderate intensity) on clinical outcomes during V-V ECMO. Before such a trial can be conducted, however, additional data are needed to inform the feasibility of the future trial.

DETAILED DESCRIPTION:
Since the inception of Extracorporeal Membrane Oxygenation (ECMO), moderate intensity titrated dose anticoagulation has been used to prevent clinically harmful thromboembolism and thrombotic mechanical complications. The impact of thromboembolic events on clinical outcomes during venovenous (V-V) extracorporeal membrane oxygenation (ECMO), however, is unclear, and complications related to bleeding are common and associated with increased morbidity and mortality. These findings have led many experts to suggest that anticoagulation strategies during V-V ECMO should be re-evaluated.

Critical illness, in general, is associated with both coagulopathy and impaired hemostasis. These problems are compounded during ECMO by the artificial interface between blood and the non-biologic surface of the circuit components, which leads to activation of the coagulation system, consumptive thrombocytopenia, fibrinolysis, and thrombin generation. The sheer stress on blood components during ECMO also lead to destruction of high-molecular-weight von Willebrand multimers, interrupting primary hemostasis.

Both bleeding and thromboembolism are common complications during ECMO. Bleeding events have been associated with poor clinical outcomes, likely mediated by an increased incidence of intracranial hemorrhage during ECMO. During intra-operative cardiopulmonary bypass and venoarterial (V-A) ECMO, ischemic strokes are a common and potentially deadly complication. During V-V ECMO, however, the majority of thromboembolic events are cannula-associated DVT and circuit thromboses requiring exchange, which are of unclear clinical significance.

Various anticoagulation strategies have been proposed to balance the risks of bleeding and thromboembolism during V-V ECMO, including high intensity anticoagulation, moderate intensity anticoagulation, and low intensity anticoagulation (the equivalent of DVT prophylaxis). Observational studies have suggested that, compared to moderate intensity anticoagulation, low intensity anticoagulation reduces transfusion requirements without affecting the incidence of thrombosis, hemorrhage, or death. In one case series of 60 patients who were treated with only low-intensity subcutaneous heparin during V-V ECMO, rates of transfusions were lower than historical controls without any effect on the rate of thrombotic events. Similarly, a recent systematic review suggested that the rates of thromboembolism and circuit thrombosis among patients managed with a moderate intensity anticoagulation strategy during V-V ECMO were comparable to the rates reported among patients managed with a less intense anticoagulation strategy.

To date, there are no randomized controlled trials comparing low intensity to moderate intensity anticoagulation during V-V ECMO. Guidelines from the Extracorporeal Life Support Organization (ELSO), the pre-eminent group for ECMO education and research, provide little guidance for the selection of anticoagulation strategy, and anticoagulation practices are highly variable across institutions. A large, multicenter, randomized trial is needed to determine the ideal strategy to anticoagulation during V-V ECMO. Before such a trial can be conducted, however, additional data are needed on the feasibility of randomizing patients to a specific anticoagulation strategy and study measurements.

To facilitate a large, multicenter randomized controlled trial comparing low intensity anticoagulation to moderate intensity anticoagulation during V-V ECMO, a pilot trial is needed to establish feasibility and the performance of the primary outcome measures.

Primary aim of the study: To demonstrate feasibility of a future large, multi-center randomized controlled trial comparing low intensity to moderate intensity anticoagulation among adults receiving V-V ECMO by demonstrating the ability to recruit and randomize participants, adhere to assigned anticoagulation strategy, and demonstrate adequate separation between groups in therapy delivered and intensity of anticoagulation achieved with the assigned anticoagulation strategies.

Secondary aim of the study: To define and estimate the frequency of the primary efficacy, primary safety, and secondary outcomes of a future large, multi-center randomized controlled trial comparing low intensity vs moderate intensity anticoagulation among adults receiving V-V ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receiving V-V ECMO
2. Patient is located in a participating unit of the Vanderbilt University Medical Center (VUMC) adult hospital.

Exclusion Criteria:

1. Patient is pregnant
2. Patient is a prisoner
3. Patient is < 18 years old
4. Patient underwent ECMO cannulation greater than 24 hours prior to screening
5. Presence of an indication for systemic anticoagulation:

   1. Ongoing receipt of systemic anticoagulation
   2. Planned administration of anticoagulation for an indication other than ECMO
   3. Presence of or plan to insert an arterial ECMO cannula
6. Presence of a contraindication to anticoagulation:

   1. Active bleeding determined by treating clinicians to make anticoagulation unsafe
   2. Major surgery or trauma less than 72 hours prior to randomization
   3. Known history of a bleeding diathesis
   4. Ongoing severe thrombocytopenia (platelet count < 30,000)
   5. History of heparin-induced thrombocytopenia (HIT)
   6. Heparin allergy
7. Positive SARS-CoV-2 test within prior 21 days or high clinical suspicion for COVID-19
8. The treating clinician determines that the patient's risks of thromboembolism or bleeding necessitate a specific approach to anticoagulation management during V-V ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Casey, MD, MSc, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Request will be reviewed by the study team and approval will be contingent upon the execution of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Aubron C, DePuydt J, Belon F, Bailey M, Schmidt M, Sheldrake J, Murphy D, Scheinkestel C, Cooper DJ, Capellier G, Pellegrino V, Pilcher D, McQuilten Z. Predictive factors of bleeding events in adults undergoing extracorporeal membrane oxygenation. Ann Intensive Care. 2016 Dec;6(1):97. doi: 10.1186/s13613-016-0196-7. Epub 2016 Oct 6. PMID 27714705
- [Background] Aubron C, Cheng AC, Pilcher D, Leong T, Magrin G, Cooper DJ, Scheinkestel C, Pellegrino V. Factors associated with outcomes of patients on extracorporeal membrane oxygenation support: a 5-year cohort study. Crit Care. 2013 Apr 18;17(2):R73. doi: 10.1186/cc12681. PMID 23594433
- [Background] Zangrillo A, Landoni G, Biondi-Zoccai G, Greco M, Greco T, Frati G, Patroniti N, Antonelli M, Pesenti A, Pappalardo F. A meta-analysis of complications and mortality of extracorporeal membrane oxygenation. Crit Care Resusc. 2013 Sep;15(3):172-8. PMID 23944202
- [Background] Combes A, Leprince P, Luyt CE, Bonnet N, Trouillet JL, Leger P, Pavie A, Chastre J. Outcomes and long-term quality-of-life of patients supported by extracorporeal membrane oxygenation for refractory cardiogenic shock. Crit Care Med. 2008 May;36(5):1404-11. doi: 10.1097/CCM.0b013e31816f7cf7. PMID 18434909
- [Background] Munshi L, Walkey A, Goligher E, Pham T, Uleryk EM, Fan E. Venovenous extracorporeal membrane oxygenation for acute respiratory distress syndrome: a systematic review and meta-analysis. Lancet Respir Med. 2019 Feb;7(2):163-172. doi: 10.1016/S2213-2600(18)30452-1. Epub 2019 Jan 11. PMID 30642776
- [Background] Murphy DA, Hockings LE, Andrews RK, Aubron C, Gardiner EE, Pellegrino VA, Davis AK. Extracorporeal membrane oxygenation-hemostatic complications. Transfus Med Rev. 2015 Apr;29(2):90-101. doi: 10.1016/j.tmrv.2014.12.001. Epub 2014 Dec 18. PMID 25595476
- [Background] Chlebowski MM, Baltagi S, Carlson M, Levy JH, Spinella PC. Clinical controversies in anticoagulation monitoring and antithrombin supplementation for ECMO. Crit Care. 2020 Jan 20;24(1):19. doi: 10.1186/s13054-020-2726-9. PMID 31959232
- [Background] Saini A, Spinella PC. Management of anticoagulation and hemostasis for pediatric extracorporeal membrane oxygenation. Clin Lab Med. 2014 Sep;34(3):655-73. doi: 10.1016/j.cll.2014.06.014. Epub 2014 Jul 24. PMID 25168949
- [Background] Doyle AJ, Hunt BJ. Current Understanding of How Extracorporeal Membrane Oxygenators Activate Haemostasis and Other Blood Components. Front Med (Lausanne). 2018 Dec 12;5:352. doi: 10.3389/fmed.2018.00352. eCollection 2018. PMID 30619862
- [Background] Tauber H, Ott H, Streif W, Weigel G, Loacker L, Fritz J, Heinz A, Velik-Salchner C. Extracorporeal membrane oxygenation induces short-term loss of high-molecular-weight von Willebrand factor multimers. Anesth Analg. 2015 Apr;120(4):730-6. doi: 10.1213/ANE.0000000000000554. PMID 25565317
- [Background] Kasirajan V, Smedira NG, McCarthy JF, Casselman F, Boparai N, McCarthy PM. Risk factors for intracranial hemorrhage in adults on extracorporeal membrane oxygenation. Eur J Cardiothorac Surg. 1999 Apr;15(4):508-14. doi: 10.1016/s1010-7940(99)00061-5. PMID 10371130
- [Background] Menaker J, Tabatabai A, Rector R, Dolly K, Kufera J, Lee E, Kon Z, Sanchez P, Pham S, Herr DL, Mazzeffi M, Rabinowitz RP, O'Connor JV, Stein DM, Scalea TM. Incidence of Cannula-Associated Deep Vein Thrombosis After Veno-Venous Extracorporeal Membrane Oxygenation. ASAIO J. 2017 Sep/Oct;63(5):588-591. doi: 10.1097/MAT.0000000000000539. PMID 28857905
- [Background] Cooper E, Burns J, Retter A, Salt G, Camporota L, Meadows CI, Langrish CC, Wyncoll D, Glover G, Ioannou N, Daly K, Barrett NA. Prevalence of Venous Thrombosis Following Venovenous Extracorporeal Membrane Oxygenation in Patients With Severe Respiratory Failure. Crit Care Med. 2015 Dec;43(12):e581-4. doi: 10.1097/CCM.0000000000001277. PMID 26308437
- [Background] Esper SA, Welsby IJ, Subramaniam K, John Wallisch W, Levy JH, Waters JH, Triulzi DJ, Hayanga JWA, Schears GJ. Adult extracorporeal membrane oxygenation: an international survey of transfusion and anticoagulation techniques. Vox Sang. 2017 Jul;112(5):443-452. doi: 10.1111/vox.12514. Epub 2017 May 3. PMID 28466601
- [Background] Krueger K, Schmutz A, Zieger B, Kalbhenn J. Venovenous Extracorporeal Membrane Oxygenation With Prophylactic Subcutaneous Anticoagulation Only: An Observational Study in More Than 60 Patients. Artif Organs. 2017 Feb;41(2):186-192. doi: 10.1111/aor.12737. Epub 2016 Jun 3. PMID 27256966
- [Background] Carter KT, Kutcher ME, Shake JG, Panos AL, Cochran RP, Creswell LL, Copeland H. Heparin-Sparing Anticoagulation Strategies Are Viable Options for Patients on Veno-Venous ECMO. J Surg Res. 2019 Nov;243:399-409. doi: 10.1016/j.jss.2019.05.050. Epub 2019 Jul 2. PMID 31277018
- [Background] Wood KL, Ayers B, Gosev I, Kumar N, Melvin AL, Barrus B, Prasad S. Venoarterial-Extracorporeal Membrane Oxygenation Without Routine Systemic Anticoagulation Decreases Adverse Events. Ann Thorac Surg. 2020 May;109(5):1458-1466. doi: 10.1016/j.athoracsur.2019.08.040. Epub 2019 Sep 26. PMID 31563493
- [Background] Olson SR, Murphree CR, Zonies D, Meyer AD, Mccarty OJT, Deloughery TG, Shatzel JJ. Thrombosis and Bleeding in Extracorporeal Membrane Oxygenation (ECMO) Without Anticoagulation: A Systematic Review. ASAIO J. 2021 Mar 1;67(3):290-296. doi: 10.1097/MAT.0000000000001230. PMID 33627603
- [Background] ELSO. ELSO Anticoagulation Guidelines. 2014.
- [Background] Bembea MM, Annich G, Rycus P, Oldenburg G, Berkowitz I, Pronovost P. Variability in anticoagulation management of patients on extracorporeal membrane oxygenation: an international survey. Pediatr Crit Care Med. 2013 Feb;14(2):e77-84. doi: 10.1097/PCC.0b013e31827127e4. PMID 23287906
- [Derived] Gannon WD, Pratt EH, Vogelsong MA, Adkisson WH, Bacchetta M, Bloom SL, Ford DJ, Guenthart BA, Landsperger JS, Qian ET, Rackley CR, Rice TW, Fielding-Singh V, Stokes JW, Stollings JL, Semler MW, Casey JD; Pragmatic Critical Care Research Group. Low-Intensity vs Moderate-Intensity Anticoagulation for Venovenous Extracorporeal Membrane Oxygenation: The Strategies for Anticoagulation During Venovenous Extracorporeal Membrane Oxygenation Pilot Trial. Chest. 2025 Sep;168(3):639-649. doi: 10.1016/j.chest.2025.02.032. Epub 2025 Mar 11. PMID 40081660

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate-intensity Anticoagulation: Patients assigned to the moderate-intensity anticoagulation group received a continuous intravenous infusion of an anticoagulant targeting a goal aPTT of 40-60 seconds or a goal anti-Xa level of 0.2 to 0.3 IU/mL. The choice of anticoagulant (e.g., heparin or bivalirudin), monitoring strategy (e.g., partial thromboplastin time or anti-Xa level), frequency of monitoring, and protocol for titrating anticoagulation to achieve goals was determined by treating clinicians and institutional protocols. The protocols used to titrate continuous infusions of anticoagulation at each center are consistent with current recommendations and protocols for patients receiving venovenous ECMO in clinical care at other centers.
- Low-intensity Anticoagulation: Patients assigned to the low-intensity anticoagulation group received intermittent subcutaneous injections of an anticoagulant at a dose used for deep venous thromboembolism prophylaxis in critically ill patients. The choice of anticoagulant (e.g. heparin or enoxaparin) and the dose used for deep venous thromboembolism prophylaxis was determined by treating clinicians and institutional protocols.
Period: Overall Study
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Intensity Anticoagulation: Moderate Intensity Anticoagulation: Participants assigned to the moderate intensity anticoagulation strategy will receive anticoagulation targeting a PTT goal of 40-60 seconds or anti-Xa level of 0.2 to 0.3 IU/mL. Choice of anticoagulant and monitoring strategy (PTT or anti-Xa level) will be at the discretion of the treating clinicians and will be prospectively recorded. Anticoagulant drips will be titrated according to institutional protocols.
  This approach to anticoagulation reflects the current approach for patients receiving V-V ECMO at Vanderbilt University Medical Center and is similar to protocols widely adopted for patients receiving V-V ECMO at other centers.
- Total: Total of all reporting groups
Arm/Group | Low Intensity Anticoagulation | Moderate Intensity Anticoagulation | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [27 to 44] | 40 [29 to 61] | 35.5 [28 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 5 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 8 | 10 | 18
  Black Non-Hispanic | 2 | 2 | 4
  Asian Non-Hispanic | 0 | 1 | 1
  Hispanic | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Bleeding Events
Description: Major bleeding event, according to the International Society on Thrombosis and Hemostasis, defined as:
  1. Fatal bleeding
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome
  3. Clinically overt bleeding associated with either a drop in hemoglobin level by at least 2.0 grams/dL or leading to transfusion of two or more units of packed red blood cells
Time Frame: From randomization to the date of death or the date 24 hours after decannulation, whichever came first, through study completion, up to 134 days.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Intensity Anticoagulation: For patients assigned to the moderate intensity anticoagulation group, clinical teams will be instructed to initiate a continuous infusion of moderate intensity anticoagulation targeting either a partial thromboplastin time (PTT) of 40-60 seconds or an Anti-Xa level of 0.2 to 0.3 IU/mL. The choice of anticoagulant and approach to dosing will be deferred to treating clinicians.
  Moderate Intensity Anticoagulation: Patients assigned to the moderate intensity anticoagulation strategy will receive anticoagulation targeting a PTT goal of 40-60 seconds or anti-Xa level of 0.2 to 0.3 IU/mL. Choice of anticoagulant and monitoring strategy (PTT or anti-Xa level) will be at the discretion of the treating clinicians and will be prospectively recorded. Anticoagulant drips will be titrated according to institutional protocols. For patients who survive to decannulation, the infusion will be stopped one hour prior to decannulation.
  This approach to anticoagulation reflects the current approach for patients receiving V-V ECMO at Vanderbilt University Medical Center and is similar to protocols widely adopted for patients receiving V-V ECMO at other centers.
Arm/Group | Low Intensity Anticoagulation | Moderate Intensity Anticoagulation
Number analyzed (Participants) | 12 | 14
Participants | 1 | 4

2. Primary Outcome: Number of Participants With Thromboembolic Events
Description: Thromboembolic event defined as:
  1. Deep venous thrombosis (DVT)
  2. Acute pulmonary embolism (PE)
  3. Intra-cardiac thrombosis
  4. Ischemic stroke
  5. Acute circuit thrombosis requiring urgent circuit exchange
  6. Acute arterial thromboembolism
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Cannula-associated Deep Vein Thrombosis
Description: Cannula-associated deep vein thrombosis, as measured by four-extremity venous ultrasounds obtained 24-72 hours following decannulation among patients who were decannulation
Time Frame: 24-72 hours after decannulation
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 7 | 5
Statistical Analysis 1: Comparison: Moderate-intensity Anticoagulation vs Low-intensity Anticoagulation; Test type: Other — Given the small sample size, simple descriptive were used. Between-group differences were performed using a Fisher exact test; p < 0.05, Fisher Exact

4. Secondary Outcome: Number of Circuit or Circuit Component Exchanges
Description: Circuit or circuit component exchange during ECMO support
Time Frame: From randomization to the date of death or decannulation, whichever came first, through study completion, up to 134 days
Measure: Number; unit: Exchanges
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Exchanges | 2 | 1

5. Secondary Outcome: New Heparin Induced Thrombocytopenia Diagnosis
Description: New diagnosis of Heparin Induced Thrombocytopenia as measured by clinically obtained serotonin release assay
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 0 | 0

6. Secondary Outcome: Lowest Platelet Count
Description: Lowest clinically obtained platelet count
Time Frame: From randomization to the the date of death or the date 24 hours after decannulation, whichever came first, through study completion, up to 134 days
Measure: Median (Inter-Quartile Range); unit: cells per mcL
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
cells per mcL | 88 [70 to 132] | 130 [115 to 170]

7. Secondary Outcome: Highest Total Bilirubin Values
Description: Highest clinically obtained total bilirubin values
Time Frame: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Low Intensity Anticoagulation | Moderate Intensity Anticoagulation
Number analyzed (Participants) | 12 | 14
mg/dL | 1.2 [0.6 to 1.4] | 0.9 [0.7 to 2.1]

8. Secondary Outcome: Highest Lactate Dehydrogenase Value
Description: Highest clinically obtained lactate dehydrogenase value
Time Frame: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
U/L | 492 [426 to 543] | 711 [320 to 941]

9. Secondary Outcome: Death Attributable to a Major Bleeding Event
Description: In-hospital mortality attributable to a major bleeding event
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 0 | 0

10. Secondary Outcome: Death Attributable to a Thromboembolic Event
Description: In-hospital mortality attributable to a thromboembolic event
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 0 | 0

11. Secondary Outcome: Ventilator-free Days
Description: Number of days alive and free from mechanical ventilation between randomization and day 28.
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
days | 54 [30 to 57] | 47 [39 to 56]

12. Secondary Outcome: ICU Length of Stay
Description: Number of days in the ICU following randomization.
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
days | 11 [6 to 20] | 15 [7 to 25]

13. Secondary Outcome: Hospital Length of Stay
Description: Number of days in the hospital following randomization
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
days | 19 [9 to 35] | 23 [14 to 45]

14. Secondary Outcome: In-hospital Mortality
Description: Death prior to hospital discharge
Time Frame: From randomization to the date of death or discharge, whichever came first, through study completion, up to 134 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 2 | 0

15. Other Pre Specified Outcome: Number of and Specific Reasons for "Missed" Enrollments
Description: Reasons for "missed" enrollments (e.g. unavailability of research staff, refusal of clinical team to allow randomization, patient refusal of informed consent)
Time Frame: From ECMO cannulation to 24 hours after ECMO cannulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
Participants | 0 | 0

16. Other Pre Specified Outcome: Duration of the Intervention Period (Days)
Description: Duration of the intervention period, defined as the time from randomization to the first of: diagnosis of a major bleeding event, diagnosis of a thromboembolic event, placement of an arterial ECMO cannula, decannulation from ECMO, or death (days)
Time Frame: From randomization to the first of decannulation or death, up to 134 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
Number analyzed (Participants) | 14 | 12
days | 4.6 [3.4 to 9.4] | 4.6 [2.6 to 6.9]

ADVERSE EVENTS:
Time Frame: From randomization to the date of death or decannulation, whichever came first, through study completion, up to 134 days
Arm/Group | Moderate-intensity Anticoagulation | Low-intensity Anticoagulation
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT04997265/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT04997265/ICF_001.pdf